CLINICAL TRIAL: NCT06220409
Title: Effect of Dance Classes on Gut Microbiota Composition, Cognitive Function, and Physical Fitness in Multiple Sclerosis Patients
Brief Title: Gut Microbiota Composition, Cognitive Function, and Physical Fitness in Multiple Sclerosis Patients
Acronym: MSDANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Principal Investigator, Viktor Bielik, prof., Comenius University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1/0260/21
Record Dates: First submitted 2024-01-09; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Sclerosis, Multiple
Keywords: Physical Activity; Gut Microbiome; Dance
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dance (Experimental): The patients persuading dance classes two times a wek for 3 months .
  Interventions: Other: Dance classes
- Passive (No Intervention): The patients engage in no structured or self-induced physical exercise or activity (sedentary individuals)
- Healthy subjects (No Intervention): The subjects engage in sports recreationally

INTERVENTIONS:
Other: Dance classes — A 12-week dance class training program two times a week for 3 months
  Arms: Dance

SUMMARY:
The evidence suggests that multiple sclerosis (MS) induces a decline in motor and cognitive function and provokes a shift in gut microbiome composition in patients. Therefore, the purpose of this study is to explore the effect of a 12-week dance class training program on the gut microbiota composition, motor function, and cognitive function of patients with MS.

The investigators will also study the following:

* The impact of organised physical activity on quality of life
* The impact of organised physical activity on body composition and metabolic parameters (e.g., insulin sensitivity, lipid profile, ect.)
* The impact of organised physical activity on physical fitness (e.g., VO2max, Power, ect.)

DETAILED DESCRIPTION:
Progressive loss of lower extremity mobility and physical function is one of the most important and well-researched effects of MS. Additionally, there is evidence that MS patients have a moderate dysbiosis in the gut microbiota structure compared to healthy subjects, whereas recent studies have demonstrated the critical role the gut microbiome plays in preserving general health, including its potential impact on neurological disorders and the immune system. Even though research is still in its early stages, the gut microbiome may have a significant impact on MS. A plethora of physical exercise strategies are available in the literature to help MS patients with fatigue, motor function, and health-related quality of life. Despite the scarcity of specific research, embracing dancing courses for MS patients has promising potential health benefits. Importantly, apart from improved physical fitness and motor function, patients with MS may also experience dancing with various other advantages, such as emotional well-being and social interaction.

Objective: This proposal aims to investigate the effects of regular physical exercise, such as dancing classes, on the health of individuals with MS. MSDANCE will investigate the impact that a dancing class training program lasting twelve weeks had on the makeup of the microbiota in the gut, as well as the motor and cognitive functioning, physical fitness, quality of life, body composition, and metabolic parameters of patients with MS. Consequently, these observations will be compared with those of healthy subjects.

Hypothesis: The investigators hypothesize that regular physical exercise (dance class training program) will improve motor and cognitive functions, with an additional positive effect on the microbial composition in patients with MS. The investigators further hypothesize the improvement in the following variables: physical fitness, quality of life, body composition, metabolic parameters, etc.

ELIGIBILITY:
Inclusion Criteria:

* patients with multiple sclerosis, diagnosed according to official diagnostic criteria according to McDonald 2010
* Consent ability and written consent
* The expanded disability status scale (EDSS) <5.5
* age 30 - 50

Exclusion Criteria:

* serious comorbidities including psychiatric diseases
* Significant cognitive impairment, clinically relevant or progressive disease (e.g., liver, kidney, cardiovascular system, respiratory tract, vascular system, brain, metabolism, thyroid) that could affect the course of the study
* Clinically relevant addiction or substance abuse disorder (defined as alcohol, drug and drug abuse)
* Nicotine consumption of > 5 cigarettes per day and no willingness to stop consumption during therapeutic fasting.
* Simultaneous participation in an interventional study or participation in an interventional study in the last two months before study inclusion
* Malignant disease
* Insufficient mental possibility of cooperation Eating disorder

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
The shift in the mean gut microbiota diversity | Change from baseline at 3 months
  Influence of the interventions on the Shannon index. The higher the index, the more diverse the species are in the habitat. The value of the Shannon-Weaver diversity index usually ranges from 1.5 to 3.5 and only rarely exceeds 4.5.
Change from baseline in the mean quantitative mobility and leg function performance | Change from baseline at 3 months
  Influence of the interventions on a time in 25-Foot Walk. The longer the duration, the worse the outcome. Normal values: less than 4 seconds; Mild impairment: 4-5.99 seconds; Moderate impairment: 6-9.99 seconds; Severe impairment: 10 seconds or more.
Change from baseline in the mean quantitative upper extremity function performance | Change from baseline at 3 months
  Influence of the interventions on a 9-hole Peg Test. The longer the duration, the worse the outcome. Values: 0 (completed without any delays) or more.
Differences in the mean quantitative maximal oxygen consumption | Changes from baseline at 3 months
  Comparison of maximal oxygen consumption (VO2max) within groups (MS pre-intervention vs. post-intervention) and between groups (healthy subjects vs. MS pre- and post-intervention). The higher the values, the better the outcome. The general ranges for VO2max in healthy adults are: Average Values: Men: 35-40 ml/kg/min, and Women: 27-31 ml/kg/min; Good Fitness Level: Men: 45-50 ml/kg/min and Women: 38-42 ml/kg/min; Excellent Fitness Level: Men: 55-60 ml/kg/min or higher, and Women: 47-52 ml/kg/min or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Bielik, prof., Principal Investigator — Faculty of Physical Education and Sport, Comenius University
Locations (1):
- Department of Biological and Medical Science, Faculty of Physical Education and Sport, Comenius University, Bratislava, Slovakia